CLINICAL TRIAL: NCT02525185
Title: Contractile Reserve in Dyssynchrony (CRID): A Novel Principle to Identify Candidates for Cardiac Resynchronization Therapy
Brief Title: Contractile Reserve in Dyssynchrony: A Novel Principle to Identify Candidates for Cardiac Resynchronization Therapy
Acronym: CRID-CRT
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Rennes University Hospital (Other); Karolinska University Hospital (Other); Onze Lieve Vrouwziekenhuis Aalst (Other)
Responsible Party: Principal Investigator, Otto Armin Smiseth, Professor, Oslo University Hospital
Other Study IDs: 2015/1022
Record Dates: First submitted 2015-08-11; First posted 2015-08-17 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure; Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Cardiomyopathies | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Diagnostic interventions; PET, MRI, cardiac ultrasound.

SUMMARY:
Cardiac resynchronisation therapy (CRT) has been documented to be a powerful treatment in patients with severe congestive heart failure. However, 30-40% of patients receiving a CRT are non-responders. In this study the investigators will use a previously validated method to estimate myocardial segment work non-invasively by speckle-tracking echocardiography and blood pressure. Furthermore, cardiac magnetic resonance imaging (CMR) with late gadolinium enhancement (LGE) will be performed in feasible subjects. The main purpose of the study is to determine if myocardial work by echocardiography in combination with viability assessment by LGE-CMR can predict response to CRT.

ELIGIBILITY:
Inclusion Criteria:

* Subject is indicated for CRT device according to European Society of Cardiology (ESC) guidelines from 2013.
* Subject is willing to sign informed consent form and is 18 years or older.

Exclusion Criteria:

* Right bundle branch block.
* Recent myocardial infarction, within 40 days prior to enrollment.
* Subject underwent coronary artery bypass graft (CABG) or valve surgery, within 90 days.
* Post heart transplantation, or is actively listed on the transplantation list, or has reasonable probability (per investigator's discretion) of undergoing transplantation in the next year
* Implanted with a LV assist device (LVAD), or has reasonable probability (per investigator's discretion) of receiving a LVAD in the next year
* Severe aortic stenosis (with a valve area of <1.0 cm2 or significant valve disease expected to be operated on within study period).
* Complex and uncorrected congenital heart disease.
* Breastfeeding women or women of child bearing potential.
* Enrolled in one or more concurrent studies that would confound the results of this study.
* Impossible to obtain LV volumes by echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are indicated for CRT device according to European Society of Cardiology (ESC) guidelines (2013).
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-09; Primary Completion 2018-07-01 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Reverse remodelling at 6 months follow-up | 6 months
  Measured by left ventricular end-systolic volume reduction of at least 15% assessed by echocardiography

SECONDARY OUTCOMES:
Reverse remodelling at 12 months follow-up | 12 months
  Measured by left ventricular end-systolic volume reduction of at least 15% assessed by echocardiography
Quality of Life Changes | 6 months
  Changes in quality of life measured by the Minnesota Living With Heart Failure Questionnaire
New York Heart Association (NYHA) Class Changes | 6 months
Heart failure hospitalizations | 12 months
Death of any cause | 5 years
Heart transplantation | 5 years
Left atrial contractile synchrony | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Otto A Smiseth, MD PhD, Principal Investigator — Oslo University Hospital; Jens-Uwe Voigt, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (2):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aalen JM, Donal E, Larsen CK, Duchenne J, Lederlin M, Cvijic M, Hubert A, Voros G, Leclercq C, Bogaert J, Hopp E, Fjeld JG, Penicka M, Linde C, Aalen OO, Kongsgard E, Galli E, Voigt JU, Smiseth OA. Imaging predictors of response to cardiac resynchronization therapy: left ventricular work asymmetry by echocardiography and septal viability by cardiac magnetic resonance. Eur Heart J. 2020 Oct 14;41(39):3813-3823. doi: 10.1093/eurheartj/ehaa603. PMID 32918449
- [Derived] Hammersboen LR, Stugaard M, Puvrez A, Larsen CK, Remme EW, Kongsgard E, Duchenne J, Galli E, Khan FH, Sletten OJ, Penicka M, Donal E, Voigt JU, Smiseth OA, Aalen JM. Mechanism and Impact of Left Atrial Dyssynchrony on Long-Term Clinical Outcome During Cardiac Resynchronization Therapy. JACC Cardiovasc Imaging. 2025 Apr;18(4):421-432. doi: 10.1016/j.jcmg.2024.09.008. Epub 2024 Nov 20. PMID 39570213
- [Derived] Larsen CK, Galli E, Duchenne J, Aalen JM, Stokke C, Fjeld JG, Degtiarova G, Claus P, Gheysens O, Saberniak J, Sirnes PA, Lyseggen E, Bogaert J, Kongsgaard E, Penicka M, Voigt JU, Donal E, Hopp E, Smiseth OA. Scar imaging in the dyssynchronous left ventricle: Accuracy of myocardial metabolism by positron emission tomography and function by echocardiographic strain. Int J Cardiol. 2023 Feb 1;372:122-129. doi: 10.1016/j.ijcard.2022.11.042. Epub 2022 Nov 29. PMID 36460211
- [Derived] Storsten P, Aalen JM, Boe E, Remme EW, Gjesdal O, Larsen CK, Andersen OS, Eriksen M, Kongsgaard E, Duchenne J, Voigt JU, Smiseth OA, Skulstad H. Mechanical Effects on Right Ventricular Function From Left Bundle Branch Block and Cardiac Resynchronization Therapy. JACC Cardiovasc Imaging. 2020 Jul;13(7):1475-1484. doi: 10.1016/j.jcmg.2019.11.016. Epub 2020 Jan 15. PMID 31954643